CLINICAL TRIAL: NCT00717912
Title: Determination of the Glycemic Index and the Insulinemic Index of a Sweetener
Brief Title: Determination of the Glycemic Index and the Insulinemic Index of a Sweetener Syrup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Routin SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SIRODEX 9708
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Healthy Volunteers
Keywords: BLOOD GLUCOSE; glycemic index; rates of digestion and absorption of food

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm 1 (Experimental): Classical sugar syrup / Classical sweetener syrup / Classical sugar syrup / Experimental sweetener syrup / Experimental sweetener syrup / Experimental sweetener syrup / Classical sugar syrup
  Interventions: Other: Experimental sweetener syrup; Other: Classical sweetener syrup; Other: Classical sugar syrup
- Arm 2 (Experimental): Experimental sweetener syrup / Experimental sweetener syrup / Classical sugar syrup / Classical sugar syrup / Classical sweetener syrup / Classical sugar syrup / Experimental sweetener syrup
  Interventions: Other: Experimental sweetener syrup; Other: Classical sweetener syrup; Other: Classical sugar syrup
- Arm 3 (Experimental): Experimental sweetener syrup / Classical sugar syrup / Experimental sweetener syrup / Classical sweetener syrup / Classical sugar syrup / Classical sugar syrup / Experimental sweetener syrup
  Interventions: Other: Experimental sweetener syrup; Other: Classical sweetener syrup; Other: Classical sugar syrup
- Arm 4 (Experimental): Experimental sweetener syrup / Experimental sweetener syrup / Experimental sweetener syrup / Classical sugar syrup / Classical sugar syrup / Classical sugar syrup / Classical sweetener syrup
  Interventions: Other: Experimental sweetener syrup; Other: Classical sweetener syrup; Other: Classical sugar syrup
- Arm 5 (Experimental): Classical sugar syrup / Experimental sweetener syrup / Classical sweetener syrup / Experimental sweetener syrup / Experimental sweetener syrup / Classical sugar syrup / Classical sugar syrup
  Interventions: Other: Experimental sweetener syrup; Other: Classical sweetener syrup; Other: Classical sugar syrup
- Arm 6 (Experimental): Experimental sweetener syrup / Experimental sweetener syrup / Experimental sweetener syrup / Classical sugar syrup / Classical sweetener syrup / Classical sugar syrup / Classical sugar syrup
  Interventions: Other: Experimental sweetener syrup; Other: Classical sweetener syrup; Other: Classical sugar syrup

INTERVENTIONS:
Other: Experimental sweetener syrup — 3 glucose and insulin responses with experimental sweetener syrup : 50 grams of digestible carbohydrate plus fiber
Other: Classical sweetener syrup — 1 glucose and insulin responses with classical sweetener syrup : 50 grams of digestible carbohydrate plus fiber
Other: Classical sugar syrup — 3 glucose and insulin responses with classical sugar syrup : 50 grams of digestible carbohydrate plus fiber

SUMMARY:
The purpose of the study is to determine the glycemic index and the insulinemic index of a sweetener syrup

DETAILED DESCRIPTION:
Glycemic index is a measure of how carbohydrate-containing foods affect blood glucose levels. All foods that contain carbohydrates, such as starchy vegetables (potatoes, corn), desserts, fruits, bread, pasta, and rice, can be tested for how they affect blood sugar levels after being eaten. Glycemic index is assessed by having one or more people eat a specific amount of a single food (usually 50 grams of digestible carbohydrate) and then measuring the change in blood sugar levels compared with the levels achieved after they have eaten a control food containing the same amount of digestible carbohydrate, such as white bread or glucose. The average change in blood sugar levels over a set period of time relative to the levels after consumption of the control food, usually white bread or glucose, is the food's glycemic index.

Insulinemic index is measure with the same methodology.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50 years
* male
* healthy volunteers
* BMI above 25 kg/m²

Exclusion Criteria:

* no medical history of hypercholesterolemia, high pressure blood, diabetes, sugar intolerance
* food allergy
* kidney deficiency
* liver troubles
* gastro-intestinal troubles
* drugs which impair sugar and lipid metabolism

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Cazaubiel, Doctor, Principal Investigator — BioFortis
Locations (1):
- Biofortis, Nantes, France

REFERENCES:
- See also: Clinical Research Organisation in Human Nutrition — http://www.biofortis.eu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Classical sugar syrup/ Classical sweetener syrup / Classical sugar syrup / Experimental sweetener syrup / Experimental sweetener syrup / Experimental sweetener syrup / Classical sugar syrup
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Started | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Each subject received the study products in different order according to the randomization list
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: participants]
  France | 6

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Index
Description: The specific measure that will be use to determine the glycemic responses is the change in blood sugar levels compared with the levels achieved after they have eaten a control food containing the same amount of digestible carbohydrate.
  Sugar syrup was used as the reference food, giving it a glycemic index value of 100 by definition. The AUC of the test food is divided by the AUC of the standard (glucose) and multiplied by 100. Low GI: 55 or less, Medium GI: 56-69, High GI: 70 and above
Time Frame: Every 48 hours (each new intervention), over a 2 hour blood glucose challenge
Measure: Mean (Standard Deviation); unit: % of GI of the glucose
Groups:
- Classical Sugar Syrup: The subjects consumed three time this product
- Experimental Sweetener Syrup: The subjects consumed three times this product
- Classical Sweetener Syrup: The subjects consumed once this product
Arm/Group | Classical Sugar Syrup | Experimental Sweetener Syrup | Classical Sweetener Syrup
Number analyzed (Participants) | 6 | 6 | 6
% of GI of the glucose | 100 (0) | 33.68 (20.28) | 12.83 (14.74)

2. Secondary Outcome: Insulinemic Index
Description: The specific measure that will be use to determine the insulinemic responses is the change in blood insuline levels compared with the levels achieved after they have eaten a control food containing the same amount of digestible carbohydrate.
  Sugar syrup was used as the reference food, giving it a insulinemic index value of 100 by definition. The AUC of the test food is divided by the AUC of the standard (glucose) and multiplied by 100. Low GI: 55 or less, Medium GI: 56-69, High GI: 70 and above
Time Frame: Every 48 hours (each new intervention), over a 2 hour blood glucose challenge
Measure: Mean (Standard Deviation); unit: % of the GI of the glucose
Groups:
- Classical Sugar Syrup; Experimental Sweetener Syrup: The subjects consumed three times this product
Arm/Group | Classical Sugar Syrup | Experimental Sweetener Syrup | Classical Sweetener Syrup
Number analyzed (Participants) | 6 | 6 | 6
% of the GI of the glucose | 100 (0) | 34.28 (16.57) | 17.38 (14.09)

ADVERSE EVENTS:
Arm/Group | Classical Sugar Syrup | Experimental Sweetener Syrup | Classical Sweetener Syrup
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 4/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Classical Sugar Syrup (N=6) | Experimental Sweetener Syrup (N=6) | Classical Sweetener Syrup (N=6)
diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days